CLINICAL TRIAL: NCT05081817
Title: Comparative Accuracy of Two Subcutaneous Continuous Glucose Monitoring Devices in Hospitalized Patients Requiring Continuous Intravenous Insulin Infusion
Brief Title: Accuracy Comparison of Two CGMs in Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Schafer Boeder, Assistant Clinical Professor, University of California, San Diego
Other Study IDs: 190045
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ICU: ICU patients on insulin drip

SUMMARY:
The purpose of the study is to determine the accuracy of two different continuous blood sugar monitoring systems in hospitalized patients by comparing them standard laboratory blood sugar testing in the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. All genders, admitted to UC San Diego Hillcrest Medical Center with an anticipated remaining length of stay of ≥24 hours
2. Age ≥18 years at the time of consent
3. Requiring standard of care intravenous insulin infusion therapy at the time of consent with an anticipated duration of intravenous insulin infusion ≥12 hours
4. Willingness to provide informed consent and follow all study procedures

Exclusion Criteria:

1. Current bleeding disorder, treatment with anticoagulants, or platelet count below 50,000/mL at enrollment
2. Lack of appropriate sites for sensor placement (sites must be free of scars, skin irritation, surgical wounds, dressings, etc.)
3. Planned magnetic resonance imaging (MRI) study within 24 hours of enrollment
4. Any other condition that, based on Investigator's judgment, would jeopardize patient safety during trial participation or would affect the study outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients requiring an insulin drip.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in glucose measurement | 5 Days
  Difference between glucose as measured by continuous glucose monitor versus laboratory

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Medical Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No